CLINICAL TRIAL: NCT04934670
Title: A Phase 3, Randomized, Open-Label, Multicenter Study, to Compare T-Guard to Ruxolitinib for the Treatment of Patients With Grade III or IV Steroid-Refractory Acute Graft-Versus-Host Disease (SR-aGVHD)
Brief Title: A Study to Compare T-Guard vs Ruxolitinib for Treatment of Steroid-Refractory Acute Graft-vs-Host Disease (BMT CTN 2002)
Acronym: 2002
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study met the protocol defined stopping boundary for Day 60 mortality when comparing mortality between the T-Guard and ruxolitinib arms
Sponsor: Xenikos (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMT CTN 2002; 5U24HL138660-02 (NIH); 2021-000343-53 (EudraCT Number); XEN-TG-005 (Other: Xenikos, BV); U10HL069294 (NIH); U24HL138660 (NIH)
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2022-04

CONDITIONS: Steroid-Refractory Acute Graft Versus Host Disease
Keywords: T-Guard; Ruxolitinib; Steroid-Refractory; GVHD; Acute GVHD; aGVHD; Grade III; Grade IV; Complete Response (CR); Transplant; Hematopoietic Stem Cell Transplant (HSCT)
MeSH Terms: conditions — Lymphoma, Follicular; Pathologic Complete Response | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at a ratio of 1:1 between the treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- T-Guard (Experimental): Participants will be administered four doses of T-Guard intravenously for a 4-hour period every other day
  Interventions: Drug: T-Guard
- Ruxolitinib (Active Comparator): Participants will take ruxolitinib twice daily for continuous daily dosing
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: T-Guard — T-Guard will be administered intravenously inpatient over 4 hours every 2 calendar days on Days 0, 2, 4, and 6, at a dose of 4mg/m2 Body Surface Area (BSA).
  Arms: T-Guard
Drug: Ruxolitinib — Ruxolitinib will be administered orally twice a day starting on Day 0 through Day 56, at a dose of 10mg. Ruxolitinib taper can be initiated starting on Day 56 for participants responding to treatment, tapering will be done according to institutional practices.
  Other Names: Jakafi; Jakavi
  Arms: Ruxolitinib

SUMMARY:
This is an open-label, randomized, Phase 3, multicenter trial, which has been designed to compare the efficacy and safety of T-Guard to ruxolitinib in patients with Grade III or IV Steroid-Refractory acute Graft-Versus-Host Disease (SR-aGVHD). The primary hypothesis is that T-Guard treatment will improve the Day 28 complete response (CR) rate in patients with Grades III and IV SR-aGVHD compared to ruxolitinib.

DETAILED DESCRIPTION:
Graft-vs-Host Disease (GVHD) is a complication that affects many hematopoietic stem cell transplant (HSCT) patients; it occurs when the new cells from a transplant attack the recipient's body. Acute GVHD (aGVHD) typically develops within the first three months after HSCT and is typically treated with steroid therapy. A significant fraction of the aGVHD population (10-50%) fail to respond to treatment and are deemed steroid-refractory (SR).

Participants that develop Grade III or IV SR aGVHD will be randomized to receive T-Guard or ruxolitinib and will be followed for approximately 180 days. Participants will be stratified by center region (US vs. Europe) and age group (at least 55 years vs. under 55). Participants randomized to the T-Guard arm will receive 4 doses administered intravenously as four 4-hour infusions, and participants randomized to the ruxolitinib arm will receive one dose administered orally twice a day. The primary analysis will include all participants that are randomized.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, patients must meet the following:

1. Patients must be at least 18.0 years of age at the time of consent.
2. Patient has undergone first allo-HSCT from any donor source or graft source. Recipients of nonmyeloablative, reduced intensity, and myeloablative conditioning regimens are eligible.
3. Patients diagnosed with Grade III/IV SR-aGVHD after allo-HSCT. SR includes aGVHD initially treated at a lower steroid dose, but must meet one of the following criteria:

   * Progressed or new organ involvement after 3 days of treatment with methylprednisolone (or equivalent) of greater than or equal to 2 mg/kg/day
   * No improvement after 7 days of primary treatment with methylprednisolone (or equivalent) of greater than or equal to 2mg/kg/day
   * Patients with visceral (GI and/or liver) plus skin aGVHD at methylprednisolone (or equivalent) initiation with improvement in skin GVHD without any improvement in visceral GVHD after 7 days of primary treatment with methylprednisolone (or equivalent) of greater than or equal to 2mg/kg/day
   * Patients who have skin GVHD alone and develop visceral aGVHD during treatment with methylprednisolone (or equivalent) of greater than or equal to 1mg/kg/day and do not improve after 3 days of greater than or equal to 2mg/kg/day Improvement or progression in organs is determined by comparing current organ staging to staging at initiation of methylprednisolone (or equivalent) treatment.
4. Patients must have evidence of myeloid engraftment (e.g., absolute neutrophil count greater than or equal to 0.5 × 109/L for 3 consecutive days if ablative therapy was previously used). Use of growth factor supplementation is allowed.
5. Patients or an impartial witness (in case the patient is capable of providing verbal consent but not capable of signing the informed consent form (ICF)) should have given written informed consent.

Exclusion Criteria:

Patients will be excluded from study entry if they meet any of the following exclusion criteria:

1. Patients who have a creatinine greater than or equal to 2mg/dL or estimated creatinine clearance less than 40 mL/min or those requiring hemodialysis.
2. Patients who have been diagnosed with active thrombotic microangiopathy (TMA), defined as meeting all the following criteria:

   * Greater than 4% schistocytes in blood (or equivalent if semiquantitative scale is used e.g., 3+ or 4+ schistocytes on peripheral blood smear)
   * De novo, prolonged or progressive thrombocytopenia (platelet count less than 50 x 109/L or 50% or greater reduction from previous counts)
   * Sudden and persistent increase in lactate dehydrogenase concentration greater than 2x the upper level of normal (ULN)
   * Decrease in hemoglobin concentration or increased transfusion requirement attributed to Coombs-negative hemolysis
   * Decrease in serum haptoglobin
3. Patients who have previously received treatment with eculizumab.
4. Patients who have previously received checkpoint inhibitors (either before or after allo-HCT).
5. Patients who have been diagnosed with overlap syndrome, that is, with any concurrent features of cGVHD.
6. Patients requiring mechanical ventilation or vasopressor support.
7. Patients who have received any systemic treatment, besides steroids, as upfront treatment of aGVHD or as treatment for SR-aGVHD. Reinstitution of previously used GVHD prophylaxis agents (e.g., tacrolimus, cyclosporin, methotrexate [MTX], MMF) or substitutes in cases with previously documented intolerance will be permitted. Previous treatment with a janus kinase (JAK) inhibitor as part of GVHD prophylaxis or treatment is not allowed.
8. Patients who have severe hypoalbuminemia, with an albumin of less than or equal to 1 g/dl.
9. Patients who have a creatine kinase (CK) level of greater than 5 times the upper limit of normal.
10. Patients with uncontrolled infections. Infections are considered controlled if appropriate therapy has been instituted and, at the time of enrollment, no signs of progression are present. Persisting fever without other signs or symptoms will not be interpreted as progressing infection. Progression of infection is defined as:

    * hemodynamic instability attributable to sepsis OR
    * new symptoms attributable to infection OR
    * worsening physical signs attributable to infection OR
    * worsening radiographic findings attributable to infection Patients with radiographic findings attributable to infection within 4 weeks prior to enrollment must have a repeat radiographic exam within one week of enrollment that documents absence of worsening.
11. Patients with evidence of relapsed, progressing, or persistent malignancy, or who have been treated for relapse after transplant, or who may require rapid immune suppression withdrawal as pre-emergent treatment of early malignancy relapse.
12. Patients with evidence of minimal residual disease requiring withdrawal of systemic immune suppression.
13. Patients with unresolved serious toxicity or complications (other than aGVHD) due to previous transplant.
14. History of sinusoidal obstruction syndrome (SOS)/veno-occlusive disease (VOD).
15. Patients with known hypersensitivity to any of the components murine monoclonal antibodies (mAb) or Recombinant Ricin Toxin A-chain (RTA).
16. Patients who have had treatment with any other investigational agent, device, or procedure within 21 days (or 5 half-lives, whichever is greater) prior to enrollment. An investigational agent is defined as medications without any known FDA or European Medicines Agency (EMA) approved indications.
17. Patients who have received more than one allo-HSCT.
18. Patients with known human immunodeficiency virus infection.
19. Patients who have a BMI greater than or equal to 35 kg/m2.
20. Patients who are taking sirolimus must discontinue prior to starting study treatment.

    The sirolimus blood level must be less than 2 ng/mL prior to starting study treatment.
21. Female patients who are pregnant, breast feeding, or, if sexually active and of childbearing potential, unwilling to use effective birth control from start of treatment until 30 days after the last study treatment.
22. Male patients who are, if sexually active and with a female partner of childbearing potential, unwilling to use effective birth control from start of treatment until 65 days after the last study treatment.
23. Patients with any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the patient; or interfere with interpretation of study data.
24. Patients whose decision to participate might be unduly influenced by perceived expectation of gain or harm by participation, such as patients in detention due to official or legal order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research; Willem Klaasen, Study Director — Xenikos, BV
Locations (48):
- United States (12):
  - University of Alabama, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Washington University St. Louis, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
- Belgium (6):
  - Site BE300, Brussels
  - Site BE301, Brussels
  - Site BE307, Ghent
  - Site BE305, Leuven
  - Site BE302, Liège
  - Site BE303, Yvoir
- Site HR320, Zagreb, Croatia
- France (10):
  - Site FR341, Angers
  - Site FR345, Créteil
  - Site FR346, La Tronche
  - Site FR355, Lille
  - SiteFR354, Nantes
  - SiteFR342, Paris
  - SiteFR348, Paris
  - Site FR356, Pierre-Bénite
  - Site FR351, Saint-Priest-en-Jarez
  - Site FR352, Toulouse
- Germany (7):
  - Site DE367, Dresden
  - Site DE364, Essen
  - Site DE371, Hanover
  - Site DE368, Heidelberg
  - Site DE360, Leipzig
  - Site DE362, Mainz
  - Site DE361, Münster
- Site IT384, Milan, Italy
- Netherlands (3):
  - Site NL461, Groningen
  - Site NL460, Maastricht
  - Site NL463, Nijmegen
- Spain (7):
  - Site ES447, Barcelona
  - Site ES446, Madrid
  - Site ES442, Salamanca
  - Site ES451, Santander
  - Site ES452, Seville
  - Site ES453, Valencia
  - Site ES454, Valencia
- Site GB483, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meyers G, Hamadani M, Martens M, Ali H, Chevallier P, Choe H, Harris AC, Holler E, van Hooren E, Klaassen W, Leifer E, van Oosterhout Y, Perez L, Pusic I, Stelljes M, van der Velden W, Ammatuna E, Beauvais D, Cornillon J, Maziarz RT, Schetelig J, Romeril J, MacMillan ML, Levine JE, Socie G. Anti-CD3/CD7 immunoconjugate (T-Guard) for severe, steroid-refractory GVHD: final report of BMT CTN 2002. Bone Marrow Transplant. 2023 Dec;58(12):1416-1418. doi: 10.1038/s41409-023-02110-4. Epub 2023 Sep 25. No abstract available. PMID 37749187
- See also: Blood and Marrow Transplant Clinical Trials Network Website — https://bmtctn.net/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T-Guard | Ruxolitinib
Started | 7 | 5
Completed | 2 | 1
Not Completed | 5 | 4
Not completed — Death | 4 | 0
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Population: A sample size of 246 participants was planned for this study with a 24-participant safety run-in. However, the study was stopped early after enrollment of 12 participants. Of these participants, 7 were randomized to T-Guard and 5 to ruxolitinib treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | T-Guard | Ruxolitinib | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Netherlands | 1 | 0 | 1
  United States | 3 | 0 | 3
  France | 3 | 3 | 6
  Germany | 0 | 2 | 2
Age 65 or above [Count of Participants; unit: Participants] | 3 | 1 | 4
Grade IV steroid-refractory aGVHD (SR-aGVHD) at randomization [Count of Participants; unit: Participants] — The severity grade of aGVHD was scored according to standard criteria (https://doi.org/10.1016/j.bbmt.2015.09.001) and ranges from Grade I to IV (with patients suffering from Grade III or IV steroid-refractory aGVHD meeting the eligibility criteria). The grading depends on the number and severity of the three target organs involved (skin, bowel and/or liver). Overall Grade I is mild, Grade II is moderate, Grade III severe and Grade IV very severe.
  Participants | 1 | 0 | 1
Hematopoietic Cell Transplantation-specific Comorbidity Index (HCT-CI) above 3 [Count of Participants; unit: Participants] | 3 | 1 | 4
Baseline serum albumin levels below 2 mg/dL [Count of Participants; unit: Participants] | 5 | 2 | 7
Absolute neutrophil count (ANC) at or below 1000/µL [Count of Participants; unit: Participants] | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR)
Description: The primary objective of this trial is to assess the rate of CR on Day 28 post-randomization in Grades III and IV SR-aGVHD patients treated with T-Guard treatment in comparison to ruxolitinib. Participants were classified as Day 28 CR if these three conditions were satisfied:
  1. Stage 0 aGVHD (no remaining symptoms) in the three target organs skin, bowel and liver, 2 . The participant is still alive at Day 28, 3 . No additional systemic treatment for aGVHD has been administered through Day 28.
Time Frame: Day 28
Population: Intention to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | T-Guard | Ruxolitinib
Number analyzed (Participants) | 7 | 5
Participants | 2 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as survival of death from any cause. The time from randomization until death from any cause will be described for each arm.
Time Frame: Day 180
Population: Participants randomized to the treatment arms were analyzed. For both treatment arms, the number of participants who died are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | T-Guard | Ruxolitinib
Number analyzed (Participants) | 7 | 5
Participants | 4 | 1

3. Secondary Outcome: Duration of Complete Response (DoCR)
Description: DoCR will be evaluated only in the set of participants who are in CR at Day 28 post-randomization. The primary definition of DoCR is the time from Day 28 until an aGVHD target organ worsens by at least 1 stage and requires a significant escalation in treatment, or death.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | T-Guard | Ruxolitinib
Number analyzed (Participants) | 7 | 5
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | T-Guard | Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 4/7 | 1/5
Serious Adverse Events (participants affected / at risk) | 5/7 | 2/5
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-Guard (N=7) | Ruxolitinib (N=5)
Enterobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infections (Infections and infestations) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Subarachnoid Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Multipel organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-Guard (N=7) | Ruxolitinib (N=5)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Factor XIII deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Conjunctival hemorrhage (Eye disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal hemorhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (5) | 0 (0)
Small intestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Edema peripheral (General disorders) | 0 (0) | 1 (1)
Physical deconditioning (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystisis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 2 (2)
Enterobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
white blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypervolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Athralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Metabolic encephalopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Azotemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vain thrombosis (Vascular disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed, which resulted in the preparation and submission to the FDA and European authorities of an abbreviated clinical study report that did not contain all the outcome measures as specified in the clinical protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT04934670/Prot_SAP_002.pdf
  • Informed Consent Form: Informed Consent to Participate in Research (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT04934670/ICF_000.pdf
  • Informed Consent Form: Pregnancy Informed Consent to Participate in Research (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04934670/ICF_001.pdf